CLINICAL TRIAL: NCT00003085
Title: Minimal Access Surgery for Pancreas Cancer: A Phase II Trial Study I: Staging of Pancreas Cancer
Brief Title: Laparoscopic Ultrasound in Diagnosing Patients With Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: CDR0000065784 (3P-94-1A); LAC-USC-3P941A; NCI-V97-1339
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Laparoscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: laparoscopy
Procedure: ultrasound imaging

SUMMARY:
RATIONALE: New diagnostic procedures, such as laparoscopic ultrasound, may improve the ability to detect pancreatic cancer and determine the extent of disease.

PURPOSE: Phase II trial to study the effectiveness of laparoscopic ultrasound in diagnosing patients with stage I or stage II pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether a comprehensive laparoscopic examination of the abdomen with laparoscopic ultrasonography improves staging of pancreatic cancer with respect to (a) better assessment (compared to CT) of the extent of localized extra pancreatic disease, (b) vascular invasion, (c) regional lymph node involvement, and (d) metastatic deposits in liver parenchyma. II. Assess whether one of the newer minimally invasive imaging techniques, laparoscopic ultrasonography, predicts vascular invasion in pancreatic cancer. III. Develop an optimal cost effective strategy for assessing resectability in pancreatic cancer.

OUTLINE: Patients who have undergone routine clinical staging (CT scan, angiogram, etc.) and who have been classified as potentially resectable undergo laparoscopy and laparoscopic ultrasound (L+LUS). At the end of the L+LUS, based on the new findings patients are reclassified as either potentially resectable or potentially unresectable. All patient then undergo definitive staging: those who have metastasis to the liver that can be pathologically confirmed by biopsy at the time of the laparoscopy are classified as unresectable and do not undergo laparotomy; all others undergo laparotomy and then are classified as resectable or unresectable. If 8 or more patients are misclassified at the time of the L+LUS, then this study is terminated.

PROJECTED ACCRUAL: There will be 50 patients accrued into this study with 25 patients in each stage. In order to accrue 50 patients, approximately 70 patients will undergo the initial routine clinical staging (CT scan, angiogram, etc.).

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histological or radiological evidence of stage I or II pancreatic cancer No evidence of metastatic disease on CT scan

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No prohibitive anesthetic risk due to cardiac disease Pulmonary: No prohibitive anesthetic risk due to respiratory disease

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: No adhesions from previous surgery that preclude laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1996-09; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dilip Parekh, MD, Study Chair — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States